CLINICAL TRIAL: NCT01219855
Title: A Randomized, Double Blind, Placebo-Controlled, Repeat Dose, Safety, Efficacy and Pharmacokinetic/Pharmacodynamic Study of CTAP101 Capsules in Subjects With Chronic Kidney Disease, Vitamin D Insufficiency and Secondary Hyperparathyroidism
Brief Title: Safety/Efficacy Study of CTAP101 in Chronic Kidney Disease Subjects With Secondary Hyperparathyroidism (SHPT)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: OPKO Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CTAP101-CL-2008
Record Dates: First submitted 2010-10-11; First posted 2010-10-13 (Estimated); Results first posted 2016-08-25 (Estimated); Last update posted 2016-08-25 (Estimated); Status verified 2014-09

CONDITIONS: Chronic Kidney Disease; Secondary Hyperparathyroidism; Vitamin D Insufficiency
Keywords: Parathyroid Diseases; Renal Insufficiency; Kidney Failure, Chronic; Hyperparathyroidism, Secondary; Vitamin D; Hyperparathyroidism; Kidney Diseases; Kidney Failure; Renal Insufficiency, Chronic
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hyperparathyroidism, Secondary; Parathyroid Diseases; Renal Insufficiency; Kidney Failure, Chronic; Hyperparathyroidism; Kidney Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Cohort 1: CTAP101 Capsules 60µg (Experimental)
  Interventions: Drug: Cohort 1 CTAP101 Capsules- 60µg
- Cohort 1: CTAP101 Capsules 90µg (Experimental)
  Interventions: Drug: Cohort 1 CTAP101 Capsules - 90µg
- Cohort 1: Sugar Capsule (Placebo Comparator)
  Interventions: Drug: Cohort 1 Matching Sugar Capsule
- Cohort 2: CTAP101 Capsules 30µg (Experimental)
  Interventions: Drug: Cohort 2 CTAP101 Capsules - 30µg
- Cohort 2: Sugar Capsule (Placebo Comparator)
  Interventions: Drug: Cohort 2 Matching Sugar Capsule

INTERVENTIONS:
Drug: Cohort 1 CTAP101 Capsules- 60µg — 60µg of CTAP101 capsules given once daily for 42 days.
  Arms: Cohort 1: CTAP101 Capsules 60µg
Drug: Cohort 1 CTAP101 Capsules - 90µg — 90µg of CTAP101 capsules given once daily for 42 days.
  Arms: Cohort 1: CTAP101 Capsules 90µg
Drug: Cohort 1 Matching Sugar Capsule — Placebo capsules given once daily for 42 days.
  Arms: Cohort 1: Sugar Capsule
Drug: Cohort 2 CTAP101 Capsules - 30µg — 30µg of CTAP101 capsules given once daily for 42 days.
  Arms: Cohort 2: CTAP101 Capsules 30µg
Drug: Cohort 2 Matching Sugar Capsule — Placebo capsules given once daily for 42 days.
  Arms: Cohort 2: Sugar Capsule

SUMMARY:
This study will investigate how the levels of a repeat dose of CTAP101 changes in the body over time (pharmacokinetics, PK) and how CTAP101 affects other mineral and hormonal balances (pharmacodynamics, PD) in patients with chronic kidney disease (CKD, vitamin D insufficiency and secondary hyperparathyroidism (SHPT).

ELIGIBILITY:
Inclusion Criteria:

1. Urinary albumin excretion of ≤3000 μg of creatinine
2. Stage 3 CKD
3. Plasma iPTH: > 70 pg/mL and < 500 pg/mL
4. Serum Ca: ≥ 8.4 mg/dL and < 10.0 mg/dL
5. Serum P: ≥ 2.0 mg/dL and < 5.0 mg/dL
6. Serum 25-hydroxyvitamin D: > 10 ng/mL and < 29 ng/mL.
7. Discontinue vitamin D use for duration of study

Exclusion Criteria:

1. History of kidney transplant or parathyroidectomy
2. Spot urine calcium:creatinine ratio > 0.2
3. Current serious illness, such as malignancy, HIV, liver disease, cardiovascular event or hepatitis
4. Currently on dialysis

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2010-10; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joel Melnick, MD, Study Director — OPKO Health, Inc.
Locations (1):
- OPKO Health, Inc, Bannockburn, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects with Stage 3 chronic kidney disease, vitamin D insufficiency and secondary parahyperthyroidism were recruited from 16 sites within the US.
Pre-assignment Details: This trial randomized 78 subjects. One subject in the 90 µg treatment arm was lost to follow-up after randomization but before receiving study drug. This subject was excluded from the Intent to Treat population (ITT).
Period: Overall Study
Arm/Group | Cohort 1: CTAP101 Capsules 60µg | Cohort 1: CTAP101 Capsules 90µg | Cohort 1: Sugar Capsule | Cohort 2: CTAP101 Capsules 30µg | Cohort 2: Sugar Capsule
Started | 17 | 17 | 17 | 13 | 14
Completed | 16 | 12 | 16 | 12 | 13
Not Completed | 1 | 5 | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Intent to treat population (excludes a single subject randomized to the 90 µg treatment arm who was lost to follow-up prior to receiving study drug)
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: CTAP101 Capsules 60µg | Cohort 1: CTAP101 Capsules 90µg | Cohort 1: Sugar Capsule | Cohort 2: CTAP101 Capsules 30µg | Cohort 2: Sugar Capsule | Total
Number analyzed (Participants) | 17 | 16 | 17 | 13 | 14 | 77
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.7 (9.20) | 64.6 (11.41) | 61.9 (17.79) | 58.2 (16.14) | 63.9 (11.47) | 63.0 (13.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 9 | 13 | 7 | 7 | 43
  Male | 10 | 7 | 4 | 6 | 7 | 34

OUTCOME MEASURES:

1. Primary Outcome: Proportion (%) of Subjects With Serum 25-hydroxyvitamin D ≥30 ng/mL (PP).
Description: The proportion of subjects in the per protocol population with serum 25-hydroxyvitamin D ≥30 ng/mL at End-of-Treatment (EOT; Week 6) in Cohorts 1 and 2 (60/90 and 30 μg groups, respectively) were compared to their corresponding placebo groups.
Time Frame: 6 weeks
Population: Per protocol
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: CTAP101 Capsules 60µg | Cohort 1: CTAP101 Capsules 90µg | Cohort 1: Sugar Capsule | Cohort 2: CTAP101 Capsules 30µg | Cohort 2: Sugar Capsule
Number analyzed (Participants) | 16 | 14 | 17 | 12 | 14
percentage of participants | 100 | 100 | 0 | 91.7 | 7.1
Statistical Analysis 1: Comparison: Cohort 1: CTAP101 Capsules 60µg vs Cohort 1: CTAP101 Capsules 90µg vs Cohort 2: CTAP101 Capsules 30µg vs Cohort 2: Sugar Capsule; Test type: Superiority or Other; p < 0.0001, Z-test cmpared 2 independ. proportions

2. Primary Outcome: Mean Percent Change From Baseline in Plasma Intact Parathyroid Hormone (iPTH) to End of Treatment (Per Protocol Population)
Description: Mean percent change from baseline in plasma intact parathyroid hormone (iPTH) from baseline to End of Treatment (EOT) in the Per Protocol population. Subjects in Cohorts 1 and 2 (dose regimens 60/90 and 30 mcg, respectively) were compared to their respective placebo groups.
Time Frame: 6 weeks
Population: Per protocol
Measure: Mean (Standard Deviation); unit: percentage of change from baseline
Arm/Group | Cohort 1: CTAP101 Capsules 60µg | Cohort 1: CTAP101 Capsules 90µg | Cohort 1: Sugar Capsule | Cohort 2: CTAP101 Capsules 30µg | Cohort 2: Sugar Capsule
Number analyzed (Participants) | 16 | 14 | 17 | 12 | 14
percentage of change from baseline | -32.77 (22.778) | -39.32 (16.243) | 20.49 (52.871) | -20.86 (21.549) | 13.18 (30.185)
Statistical Analysis 1: Comparison: Cohort 2: CTAP101 Capsules 30µg vs Cohort 2: Sugar Capsule; Test type: Superiority or Other; p < 0.01, Mixed effect model

3. Secondary Outcome: Change From Baseline in Serum 25-hydroxyvitamin D at Week 6
Description: Mean absolute change from baseline in serum total 25-hydroxyvitamin D to end of treatment (EOT)
Time Frame: Baseline to End of Treatment (6 weeks)
Population: Per protocol population
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 1: CTAP101 Capsules 60µg | Cohort 1: CTAP101 Capsules 90µg | Cohort 1: Sugar Capsule | Cohort 2: CTAP101 Capsules 30µg | Cohort 2: Sugar Capsule
Number analyzed (Participants) | 16 | 14 | 17 | 12 | 14
ng/mL | 43.25 (16.519) | 63.69 (17.826) | -0.65 (2.502) | 16.22 (6.005) | -1.89 (4.913)
Statistical Analysis 1: Comparison: Cohort 1: CTAP101 Capsules 60µg vs Cohort 1: CTAP101 Capsules 90µg vs Cohort 1: Sugar Capsule vs Cohort 2: CTAP101 Capsules 30µg vs Cohort 2: Sugar Capsule; Test type: Superiority or Other; p < 0.0001, Mixed effect model
Statistical Analysis 2: Comparison: Cohort 2: CTAP101 Capsules 30µg vs Cohort 2: Sugar Capsule; Test type: Superiority or Other; p < 0.01, Mixed effect model

4. Secondary Outcome: Percent Change From Baseline in Serum 25-hydroxyvitamin D at End of Treatment (EOT, Week 6) in the Per Protocol Population
Description: Mean percent change from baseline in serum 25-hydroxyvitamin D at End of Treatment (EOT, week 6) in the per protocol population. Subjects in Cohorts 1 and 2 (dose regimens of 60/90 and 30 mcg, respectively) were compared versus their corresponding placebo groups.
Time Frame: Baseline to End of Treatment (6 weeks)
Population: Per protocol population
Measure: Mean (Standard Deviation); unit: percentage of change from baseline
Arm/Group | Cohort 1: CTAP101 Capsules 60µg | Cohort 1: CTAP101 Capsules 90µg | Cohort 1: Sugar Capsule | Cohort 2: CTAP101 Capsules 30µg | Cohort 2: Sugar Capsule
Number analyzed (Participants) | 16 | 14 | 17 | 12 | 14
percentage of change from baseline | 187.64 (74.251) | 313.12 (101.592) | -2.67 (13.069) | 90.90 (62.189) | -7.22 (20.599)
Statistical Analysis 1: Comparison: Cohort 1: CTAP101 Capsules 60µg vs Cohort 1: CTAP101 Capsules 90µg vs Cohort 1: Sugar Capsule vs Cohort 2: CTAP101 Capsules 30µg vs Cohort 2: Sugar Capsule; Test type: Superiority or Other; p < 0.0001, Mixed effect model

5. Secondary Outcome: Proportion of Subjects With Reduction of Intact Parathyroid Hormone (iPTH) of at Least 30% at Week 6
Description: Proportion of subjects with at least 30% reduction in plasma intact parathyroid hormone (iPTH) and/or mean iPTH reduction to 70 pg/mL or less at End of Treatment (EOT)
Time Frame: Baseline to End of Treatment (6 weeks)
Population: Per protocol
Measure: Number; unit: participants
Arm/Group | Cohort 1: CTAP101 Capsules 60µg | Cohort 1: CTAP101 Capsules 90µg | Cohort 1: Sugar Capsule | Cohort 2: CTAP101 Capsules 30µg | Cohort 2: Sugar Capsule
Number analyzed (Participants) | 16 | 14 | 17 | 12 | 14
participants | 11 | 9 | 2 | 5 | 0
Statistical Analysis 1: Comparison: Cohort 1: CTAP101 Capsules 60µg vs Cohort 1: CTAP101 Capsules 90µg vs Cohort 1: Sugar Capsule vs Cohort 2: CTAP101 Capsules 30µg vs Cohort 2: Sugar Capsule; Test type: Superiority or Other; p < 0.05, Z-test compared 2 independ. proportions

6. Secondary Outcome: Proportion of Subjects With Reduction of Intact Parathyroid Hormone (iPTH) of at Least 20% at Week 6
Description: Proportion of subjects with at least 20% reduction in plasma intact parathyroid hormone (iPTH) and/or mean iPTH reduction to 70 pg/mL or less at End of Treatment (EOT)
Time Frame: Baseline to End of Treatment (6 weeks)
Population: Per protocol population
Measure: Number; unit: participants
Arm/Group | Cohort 1: CTAP101 Capsules 60µg | Cohort 1: CTAP101 Capsules 90µg | Cohort 1: Sugar Capsule | Cohort 2: CTAP101 Capsules 30µg | Cohort 2: Sugar Capsule
Number analyzed (Participants) | 16 | 14 | 17 | 12 | 14
participants | 12 | 13 | 2 | 5 | 1
Statistical Analysis 1: Comparison: Cohort 1: CTAP101 Capsules 60µg vs Cohort 1: CTAP101 Capsules 90µg vs Cohort 1: Sugar Capsule; The proportion of subjects achieving a ≥20% decrease in plasma iPTH at EOT was greater in the CTAP101 Capsules 60 and 90 μg groups compared to the corresponding placebo group; Test type: Superiority or Other; p < 0.001, Z-test compared 2 independ. proportions

ADVERSE EVENTS:
Time Frame: 12 weeks (6 week treatment period, followed by 6 week follow-up period)
Groups:
- Cohorts 1,2: Sugar Capsule: Cohort 1 Matching Sugar Capsule: Placebo capsules given once daily for 42 days.
Arm/Group | Cohorts 1,2: Sugar Capsule | Cohort 2: CTAP101 Capsules 30µg | Cohort 1: CTAP101 Capsules 60µg | Cohort 1: CTAP101 Capsules 90µg
Serious Adverse Events (participants affected / at risk) | 1/31 | 1/13 | 1/17 | 1/16
Other Adverse Events (participants affected / at risk) | 22/31 | 8/13 | 12/17 | 10/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohorts 1,2: Sugar Capsule (N=31) | Cohort 2: CTAP101 Capsules 30µg (N=13) | Cohort 1: CTAP101 Capsules 60µg (N=17) | Cohort 1: CTAP101 Capsules 90µg (N=16)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Unrelated to study drug
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) — Unrelated to study drug
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Unrelated to study drug
Angioplasty (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Unrelated to study drug
Hypoglycaemia (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Unrelated to study drug
Acute prerenal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Unrelated to study drug
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Unrelated to study drug
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohorts 1,2: Sugar Capsule (N=31) | Cohort 2: CTAP101 Capsules 30µg (N=13) | Cohort 1: CTAP101 Capsules 60µg (N=17) | Cohort 1: CTAP101 Capsules 90µg (N=16)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemia (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Frequent bowel movements (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Tooth impacted (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Impaired healing (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 3 (3) | 0 (0) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 0 (0) | 2 (2)
Fractured sacrum (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Patella fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood 25-hydroxycholecalciferol increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Body temperature increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vitamin D increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hyperphosphatemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Magnesium deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Joint warmth (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1) | 2 (2)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Tearfulness (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Telangiectasia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthma prophylaxis (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1) | 2 (2)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vessel puncture site haematoma (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flank pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eschar (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sunburn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood uric acid increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypogeusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sensory loss (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depressed mood (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Restlessness (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less